CLINICAL TRIAL: NCT06742164
Title: Role of Ivabradine for Heart Rate Control in Management of Patients With Sepsis and Septic Shock
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, Assistant Professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ms 719/2023
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Heart Rhythm Disorder
MeSH Terms: interventions — Ivabradine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients received Ivabradine (Active Comparator)
  Interventions: Drug: Ivabradine 5mg Tab
- Patients didn't receive Ivabradine . (Sham Comparator)
  Interventions: Drug: control

INTERVENTIONS:
Drug: Ivabradine 5mg Tab — Ivabradine (5 mg twice daily) orally or via nasogastric tube
  Arms: Patients received Ivabradine
Drug: control — Patients didn't receive Ivabradine .
  Arms: Patients didn't receive Ivabradine .

SUMMARY:
Tachycardia is associated with excess mortality during septic shock. This may be related to the increase in cardiac metabolic demand, impaired cardiac diastolic function and less effect of administered exogenous catecholamines.

In this study, we evaluate the effect of enteral Ivabradine on outcome of septic patients regarding need for vasopressor therapy, mechanical ventilation, renal replacement therapy, length of ICU stay and in-hospital mortality.

DETAILED DESCRIPTION:
All patients will be subjected to:

1. Thorough history taking:

   * Demographic data: age, sex and residence.
   * Clinical presentation (fever, hypotension , tachycardia , tachypnea and anuria) .
   * Family history of immunodeficiency disease
   * History of recurrent
2. Clinical examination:

   * Vital signs: heart rate (HR) , blood pressure (BP), and temperature.
   * Abdominal examination .
   * Detect septic focus .
   * Urine out put .
   * Follow up until discharge from ICU.
3. Laboratory investigations:

All patient will be screened with :

* Kidney function test .
* Liver function test.
* Total leukocyticcount was assessed immediately after admission to ICU and then every other day
* C-reactive protien was assessed immediately after admission to ICU and then every other day
* Broad-spectrum antibiotic and then according to cultures and sensitivity.
* Radiological investigation .
* Abdominal ultrasound.
* ECG.
* Echocardiography.

Study tools and procedures:

Epidemiological, demographic, clinical, laboratory, treatment, and outcome data will be obtained from medical records using a standardized data collection form.

Data will be obtained by Randomized controlled clinical trial (RCT) of medical records after, the study methodology reviewed and approved by the Research Review Board of Alhelal hospital (Intensive care unit), Faculty of medicine, Ain Shams University hospitals (Intensive care unit) .

The point of enrolment after initial haemodynamic stabilisation was taken as time 0. The following data sets were recorded at the specified time intervals.

An arterial line and central venous catheter were inserted in all patients for invasive blood pressure and central venous pressure monitoring. The point of enrolment after initial haemodynamic stabilisation was taken as time 0.

If the heart rate was less than 70 beats /min. the dose was omitted. The initial mangement of patients with sepsis and septic shock is summarised on three pillars of therapy.

Stabilization of haemodynamics with target mean arterial blood pressure at 65 mmHg for most patients, begain to rapidly administer 30ml/kg balanced crystalloid within 3 hours for hypotension or lactate ≥ 4mmol/L , Apply vasopressor if hypotensive during or after fluid resuscitation (The vasopressor of choice in septic shock is noradrenaline) , Hydrocortisone 100-200 mg/day is added In patients with refractory hypotension Obtain blood cultures before administration antibiotics. Control source of sepsis. Patients in group (A)were administered 5 mg ivabradine ( orally or crushed and injected through the enteral feeding tube every 12 hours.Heart rate was assessed prior to each dose.

Group (B): Patients didn't receive Ivabradine .

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven or suspected site of infection.
* Patients sepsis (acute organ dysfunction secondary to documented or suspected infection)
* Patients with septic shock (defined as hypotension unresponsive to fluid resuscitation and requiring vasopressor treatment to maintain adequate blood pressure) for at least 6 hours and less than 24 hours.
* Patients with sinus rhythm with heart rate ≥ 95 bpm at time of randomization. Informed consent obtained in accordance with local regulations.

Exclusion Criteria:

* Cardiac arrhythmia, conduction disorder, sinus syndrome ("sick sinus syndrome"), atrial fibrillation and heart block.
* Cardiogenic shock or acute heart failure, without proven or suspected infection.
* Acute coronary syndrome.
* Refractory shock with systolic arterial pressure <90 mm Hg despite the use of high doses of vasopressors.
* Co-treatment with drugs inducing bradycardia.
* Patients with pacemakers.
* Known pregnancy, breast-feeding, women with of childbearing potential will be tested for pregnancy and excluded if pregnant.
* Known allergy to Ivabradine
* Severe renal failure (creatinine clearance <15 ml/min) or hepatic failure (prothrombin time <20%)
* Tachycardia due to hyperthyroidism, pheochromocytoma or severe anemia (<7 g/dl)
* Enteral feeding impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
the percentage of patients with heart rate reduction of at least 10 beats/min | after 72 hours of treatment

SECONDARY OUTCOMES:
Mean heart rate | 72 hours of treatment
Mean arterial blood pressure | 72 hours of treatment
percentage of patients needed vasopressor | 72 hours of treatment